CLINICAL TRIAL: NCT03574844
Title: Randomized, Double-blind, Placebo-controlled Clinical Study Evaluating the Effect of Oral Probiotic Yeast on the Composition of the Vaginal Microbiota in Healthy Women
Brief Title: Effect of Oral Probiotic Yeast on the Composition of the Vaginal Microbiota in Healthy Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lesaffre International (Industry)
Collaborators: Biofortis Mérieux Nutriscience (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017-A02709-44
Record Dates: First submitted 2018-06-11; First posted 2018-07-02 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2018-06

CONDITIONS: Vaginal Health

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, 3 parallel-arms, pilot clinical study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Saccharomyces cerevisiae, dose 500 (Experimental): Saccharomyces cerevisiae CNCM I-3856, 500 mg per day (2 capsules), for 4 weeks
  Interventions: Dietary Supplement: Saccharomyces cerevisiae, dose 500
- Saccharomyces cerevisiae, dose 1000 (Experimental): Saccharomyces cerevisiae CNCM I-3856, 1 g per day (2 capsules), for 4 weeks
  Interventions: Dietary Supplement: Saccharomyces cerevisiae, dose 1000
- Placebo (Placebo Comparator): Maize starch and magnesium stearate, 1 g per day (2 capsules), for 4 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Saccharomyces cerevisiae, dose 500 — Experimental arm
  Arms: Saccharomyces cerevisiae, dose 500
Dietary Supplement: Saccharomyces cerevisiae, dose 1000 — Experimental arm
  Arms: Saccharomyces cerevisiae, dose 1000
Dietary Supplement: Placebo — Placebo comparator arm
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the impact of oral consumption of the probiotic yeast CNCM I-3856 on healthy vaginal microbiota

ELIGIBILITY:
Inclusion Criteria:

* Caucasian or Asian women,
* With regular menstrual cycles, assessed as 28 days ± 3 days,
* With a normal vaginal flora : Nugent score ≤ 3,
* With the same efficient contraception method since at least 3 months before the start of the study, and accepting to maintain this program over the study. Authorized contraception methods: hormonal contraception (pill, patch, implant and intrauterine device), tubal ligation, ESSURE system and copper intrauterine device (without hormone),
* Agreeing to keep unchanged her intimate hygiene rules during the all duration of the study (same stable intimate hygiene habits since at least 3 months before the start of the study),
* Good general and mental health compatible with the study participation and allowing to be followed in ambulatory way according to the investigator opinion: no clinically significant and relevant abnormalities of medical history or physical examination;
* Having stable life habits since at least 3 months and accepting to maintain them stable during the study (dietary habits, tobacco and alcohol consumptions, physical activity and sexual activity),
* Tobacco consumption ≤ 10 cigarettes per day,
* Able and willing to participate to the study by complying with the protocol procedures (especially concerning study product consumption and biological samples collections), as evidenced by her dated and signed informed consent form,
* Affiliated with a social security scheme,
* Agreeing to be registered on the national file of volunteers participating in biomedical research.

Exclusion Criteria:

* Having hypersensitivity history to one of the ingredients of the study products,
* Suffering from a metabolic disorder such as diabetes, uncontrolled thyroidal trouble or other uncontrolled metabolic disorder,
* Suffering from a severe chronic disease (e.g. cancer, renal failure, hepatic or biliary disorders ongoing, chronic inflammatory digestive disease, arthritis, chronic respiratory trouble, chronic gastro-intestinal disorder, cardiac disease, immunodeficiency…) or diseases found to be inconsistent with the conduct of the study by the investigator (controlled arterial hypertension accepted),
* Suffering from Sexually Transmitted Infection (STI) or Disease (STD) such as HIV (Human Immunodeficiency Virus), B and C hepatitis, HPV (Human PapillomaVirus), Chlamydia infection, syphilis, gonorrhea, genital herpes, etc,
* Currently suffering or having suffer from bacterial, fungal, parasitic or viral infection of the uro-gynecological sphere (vaginitis, cystitis, cervix infection…), treated or not, in the 6 months previous to the study start,
* Having medical history or current pathology which could affect the study results or expose the subject to an additional risk according to the investigator,
* Currently pregnant, or lactating, intending to be pregnant within 2 months ahead or pregnancy and/or breastfeeding finished since less than 3 months,
* Ongoing symptoms of vaginal and/or urinary infection (belong to symptoms questionnaire) at the moment of the V0 and V1 visits,
* Recent history of radiotherapy (less than 6 months),
* Menopausal or pre-menopausal,
* With menstruation which usually lasts more than 7 days,
* Under chronic treatment with corticosteroids and/or immune modulator (immunostimulant, immunosuppressant…) or last intake within 3 months before the start of the study,
* Currently under medication or dietary supplement, oral or local, which could affect study parameters: antibiotic, antifungal, probiotic, prebiotic, symbiotic, phytoestrogens, etc, or stopped within a too short time window before study start (less than 4 weeks) ,

  .- Having a lifestyle deemed incompatible with the study according to the investigator (specific diet (vegetarian, vegan, hypocolaric…), alcohol consumption > 2 glasses / day, physical activity > 10 hours / week…),
* With a personal history of anorexia nervosa, bulimia or significant eating disorders according to the investigator,
* Planning to travel for a long time during the study duration or not able to be contacted for emergency reason during the study available,
* Presenting a psychological or linguistic incapacity to understand and sign the informed consent,
* Participating in another clinical trial or in exclusion period from a previous clinical trial,
* Having received, during the last 12 months, countervailing indemnities for clinical trial higher or equal to 4500 Euros,
* Under legal protection (guardianship, wardship) or deprived from her rights following judicial or administrative decision.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
S cerevisiae transfer from the gut to the vagina | Day 28
  Proportion of subjects presenting the yeast strain S cerevisiae CNCM I-3856 (presence) in their vaginal microbiota after a 4-week daily supplementation

SECONDARY OUTCOMES:
S cerevisiae transfer from the gut to the vagina | Day 7, Day 14, Day 21, Day 42
  Proportion of subjects presenting the yeast strain S cerevisiae CNCM I-3856 (presence) in their vaginal microbiota after 1, 2 or 3-week daily supplementation and after a 2-week observation period without supplementation
Quantification of S cerevisiae in the vagina | Day 7, Day 14, Day 21, Day 28, Day 42
  Value at Day 7, 14, 21, 28, 42 and change Day 42 - Day 28 of S cerevisiae CNCM I-3856 (CFU/ sample) in the vaginal microbiota
Impact on 4 predominant Lactobacilli species | Day 7, Day 14, Day 21, Day 28, Day 42
  Changes of 4 dominant Lactobacilli species (number of copies per sample) by comparison of the 3 groups at each time change
Association between intestinal and vaginal microbiota for the presence of S cerevisiae CNCM I-3856 | Day 7, Day 14, Day 21, Day 28, Day 42
  Evaluation of the presence of S cerevisiae CNCM I-3856 in the vaginal microbiota considering its presence in the intestinal microbiota in each active group.
Correlation between the quantity of S cerevisiae CNCM I-3856 (CFU/sample) in the intestinal microbiota and vaginal microbiota | Day 7, Day 14, Day 21, Day 28, Day 42
  Correlation between the quantity of S cerevisiae CNCM I-3856 (CFU/sample) in the intestinal microbiota and vaginal microbiota in each active group.
Presence of Candida albicans in the vaginal microbiota | Day 7, Day 14, Day 21, Day 28, Day 42
  In each group, at each time point according to Day 0 and at Day 42 according to Day 28
Evolution of the presence of Candida albicans in the vaginal microbiota | Day 7, Day 14, Day 21, Day 28, Day 42
  Changes of Candida albicans (CFU/samples) in the vaginal microbiota

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis Mérieux Nutriscience, Saint-Herblain, France